CLINICAL TRIAL: NCT01078298
Title: A Phase 4 12-week, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating The Safety And Efficacy Of Varenicline Tartrate (CP-526,555) 1mg BID For Smoking Cessation In Subjects With Depression
Brief Title: Safety And Efficacy Of 12 Weeks Of Varenicline For Smoking Cessation In Smokers With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051122
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-03

CONDITIONS: Smoking Cessation; Depression
Keywords: smoking; smoking cessation; smoking cessation in depressed subjects
MeSH Terms: conditions — Smoking Cessation; Depression; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Experimental)
  Interventions: Drug: varenicline
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — varenicline tablets titrated to 1 mg BID during 1st week and then 1 mg BID for 11 weeks
  Other Names: Champix/Chantix
  Arms: varenicline
Drug: placebo — placebo tablets matched in appearance and dosage to varenicline tablets
  Arms: placebo

SUMMARY:
Patients with depression tend to have a higher prevalence of smoking as well as increased severity of nicotine dependence. Phase 2 and Phase 3 varenicline clinical trials that demonstrated its efficacy and tolerability have not included subjects with depression. This smoking cessation study focuses on the depressed population and will assess the efficacy and safety of varenicline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female cigarette smokers, 18-75 years, motivated to stop smoking and considered suitable for a smoking cessation attempt
* Smoked an average of at least 10 cigarettes per day during past year and over past month, and exhaled carbon monoxide (CO) > 10 ppm at screening
* Current or past diagnosis of MDD without psychotic features, either single or recurrent, using DSM IV TR based on clinical assessment and confirmed by SCID and at least one of the following:
* On stable antidepressant treatment for MDD (stable dose for at least 2 months)
* Major depressive episode, using DSM IV TR, in the past 2 years successfully treated

Exclusion Criteria:

* Current or past diagnosis of dementia, schizophrenia, schizoaffective disorder, or other psychotic disorder, bipolar I disorder, bipolar II disorder.
* Subjects with antisocial, schizotypal, or any other personality disorder severe enough to compromise the subject's ability to comply with the study requirements..
* Current use of either bupropion or nortryptiline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (16):
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - Behavioral Health and Wellness Program, University of Colorado Denver, Aurora, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Emerald Coast Mood & Memory, PA, Fort Walton Beach, Florida
  - Clinical Neuroscience Solutions Incorporated, Jacksonville, Florida
  - Clinical Neuroscience Solutions Incorporated, Orlando, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Vince and Associates Clinical Research, Overland, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - NorthCoast Clinical Trials Inc., Beachwood, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - CRI Worldwide LLC, Philadelphia, Pennsylvania
  - Clinical Trials of Memphis, Bartlett, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Research Clinic, Ltd., Houston, Texas
- Bosnia and Herzegovina (2):
  - Psychiatric Clinic, Clinical Center Banja Luka, Banja Luka
  - Clinic of Psychiatry, Clinical Center University of Sarajevo, Sarajevo
- Croatia (2):
  - "Poliklinika Neuron" - Croatian Institute for Brain Research, Zagreb
  - Psychiatric Hospital Vrapce, Zagreb
- Germany (3):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Ludwig Maximilians-Universitaet Muenchen, München
  - Universitaetsklinik Tuebingen, Klinik fuer Psychiatrie und Psychotherapie, Tübingen
- Hungary (6):
  - Fovarosi Onkormanyzat Nyiro Gyula Korhaz, II. Pszichiatriai Osztaly, Budapest
  - Processus Kft., Varoskapu Rendelo, Budapest
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza, Pszichiatriai Osztaly, Gyula
  - Varosi Egeszsegugyi Kozpont, Kunszentmárton
  - Donatella 99 Bt., Szentes
  - Fejer Megyei Szent Gyorgy Korhaz, Pszichiatriai Osztaly, Székesfehérvár
- Romania (3):
  - Spitalul Clinic de Psihiatrie Socola, sectia VII, Iași, Iaşi
  - Spitalul Psihiatrie "Prof. Dr. Al. Obregia", Bucharest, Sector 4
  - Spitalul Clinic de Psihiatrie Prof. Dr. Al. Obregia, sectia 2, Bucharest
- Russia (4):
  - Federal State Institution Moscow Scientific Research Institute of Psychiatry of Roszdrav, Moscow
  - Institution of Russian Academy of Medical Sciences Mental Health Research Center, Moscow
  - Moscow State Healthcare Institution Clinical Mental Hospital No 12, Moscow
  - St-Petersburg State Healthcare Institution St. Nicholas Mental Hospital, Saint Petersburg
- Spain (4):
  - Hospital de La Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital General de La Vall D'Hebron, Barcelona, Barcelona
  - Centro de Salud Mental Ii "La Corredoria", Oviedo, Principality of Asturias
  - Centro de Salud Torrero La Paz, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Anthenelli RM, Morris C, Ramey TS, Dubrava SJ, Tsilkos K, Russ C, Yunis C. Effects of varenicline on smoking cessation in adults with stably treated current or past major depression: a randomized trial. Ann Intern Med. 2013 Sep 17;159(6):390-400. doi: 10.7326/0003-4819-159-6-201309170-00005. PMID 24042367
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051122&StudyName=Safety%20And%20Efficacy%20Of%2012%20Weeks%20Of%20Varenicline%20For%20Smoking%20Cessation%20In%20Smokers%20With%20Depression%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Varenicline 0.5 milligram (mg) tablet given orally once daily up to Day 3 followed by varenicline 0.5 mg tablet orally twice daily up to Day 7 and then varenicline 1 mg tablet given orally twice daily up to Week 12. Participants were followed-up for additional 40 weeks post-treatment.
- Placebo: Placebo matched to varenicline 0.5 mg tablet orally once daily up to Day 3 followed by placebo matched to varenicline 0.5 mg tablet orally twice daily up to Day 7 and then placebo matched to varenicline 1 mg tablet orally twice daily up to Week 12. Participants were followed-up for additional 40 weeks post-treatment.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 256 | 269
Completed | 175 | 179
Not Completed | 81 | 90
Not completed — Lost to Follow-up | 12 | 13
Not completed — Withdrawal by Subject | 31 | 33
Not completed — Protocol Violation | 6 | 6
Not completed — Adverse Event | 6 | 5
Not completed — Death | 2 | 0
Not completed — Did not meet entrance criteria | 0 | 1
Not completed — Other | 24 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 256 | 269 | 525
Age, Customized [Number; unit: participants]
  18 to 44 years | 106 | 98 | 204
  45 to 64 years | 146 | 160 | 306
  Greater than or equal to 65 years | 4 | 11 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 170 | 329
  Male | 97 | 99 | 196

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Four-Week Continuous Quit Rate (CQR)
Description: Percentage of participants who reported no use of nicotine-containing products by answering "No" to the nicotine use inventory (NUI) questions: 'Has the participant smoked cigarettes' and 'Has the participant used other nicotine-containing products' in the last 7 days (Week 9) or since last study visit (Week 9 through 12) confirmed by a measurement of an end-expiratory exhaled carbon monoxide (CO) measurement less than or equal to 10 parts per million (ppm).
Time Frame: Week 9 through Week 12
Population: All participants analysis set included all the participants who were randomized and took at least one dose of randomized study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
Percentage of participants | 35.9 | 15.6
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Odds Ratios and p-values were obtained from a logistic regression model including the main effects of treatment, pooled center and cohort; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.35, 95% CI 2-sided [2.16 to 5.21]

2. Secondary Outcome: Percentage of Participants With Continuous Abstinence Rate (CAR)
Description: Percentage of participants who remained abstinent from the period defined as start of the primary endpoint (Week 9) through Week 24 and the end of follow-up (Week 52) by reporting no use of nicotine-containing products confirmed by a measurement of an end-expiratory exhaled CO measurement less than or equal to 10 ppm.
Time Frame: Week 9 through Week 24, Week 9 through Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
Percentage of participants
  Week 9 through Week 24 | 25.0 | 12.3
  Week 9 through Week 52 | 20.3 | 10.4
Statistical Analysis 1: Comparison: Varenicline vs Placebo; For Week 9 through 24, odds ratio and p-value were calculated from logistic regression model including the main effects of treatment, pooled center and cohort; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.56 to 4.10]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; For Week 9 through 52, odds ratio and p-value were calculated from logistic regression model including the main effects of treatment, pooled center and cohort; Test type: Superiority or Other; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.40 to 3.98]

3. Secondary Outcome: Number of Participants With 7-day Point Prevalence (PP) of Abstinence
Description: Number of participants reporting no use of nicotine-containing products in the last 7 days confirmed by a measurement of an end-expiratory exhaled CO measurement less than or equal to 10 ppm.
Time Frame: Weeks 12, 24, 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
participants
  Week 12 | 118 | 54
  Week 24 | 80 | 49
  Week 52 | 73 | 47
Statistical Analysis 1: Comparison: Varenicline vs Placebo; For Week 12, odds ratio and p-values were obtained from a logistic regression model including the main effects of treatment, pooled center and cohort; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.82, 95% CI 2-sided [2.53 to 5.78]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; For Week 24, odds ratio and p-values were obtained from a logistic regression model including the main effects of treatment, pooled center and cohort; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.40 to 3.33]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; For Week 52, odds ratio and p-values were obtained from a logistic regression model including the main effects of treatment, pooled center and cohort; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.28 to 3.08]

4. Secondary Outcome: Number of Participants With 4-Week Point Prevalence (PP) of Abstinence
Description: Number of participants at Week 52 visit reporting no smoking and no use of other tobacco products in the last 4 weeks confirmed by a measurement of an end-expiratory exhaled CO measurement less than or equal to 10 ppm.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
participants | 70 | 45
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0027, Regression, Logistic; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.26 to 3.08]

5. Other Pre Specified Outcome: Number of Participants With Adverse Events (Including Solicited Neuropsychiatric Adverse Events)
Description: Adverse Event (AE):any untoward medical occurrence attributed to study drug in participant who received study drug.SAE:AE causing:death;initial/prolonged inpatient hospitalization;life-threatening experience(immediate risk of dying);persistent/significant disability/incapacity;congenital anomaly.Solicited AEs collected by semi-structured neuropsychiatric AEs interview inquiring about AEs:delusions,hallucinations,paranoia,psychosis,mania,panic,agitation,hostility,aggression,homicidal ideation. If participant had positive response,investigator determined if it met AE criteria.
Time Frame: Baseline up to Week 16
Population: Safety analysis population included all participants who took at least 1 dose of randomized study medication, including partial doses, and had a safety measurement.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
participants | 185 | 180

6. Other Pre Specified Outcome: Number of Participants With Categorical Scores on Clinical Global Impression - Improvement (CGI-I)
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement from baseline is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 16, 24, 32, 40, 52
Population: Safety analysis population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' is signifying those participants who were evaluated for this measure at the time point for each group respectively.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 250 | 263
participants
  Week 1: very much improved(n=250,263) | 1 | 2
  Week 1: much improved(n=250,263) | 12 | 6
  Week 1: minimally improved(n=250,263) | 31 | 21
  Week 1: no change(n=250,263) | 189 | 222
  Week 1: minimally worse(n=250,263) | 16 | 11
  Week 1: much worse(n=250,263) | 1 | 1
  Week 2: very much improved(n=244,255) | 2 | 1
  Week 2: much improved(n=244,255) | 18 | 12
  Week 2: minimally improved(n=244,255) | 33 | 38
  Week 2: no change(n=244,255) | 159 | 181
  Week 2: minimally worse(n=244,255) | 27 | 21
  Week 2: much worse(n=244,255) | 5 | 2
  Week 3: very much improved(n=241,248) | 10 | 4
  Week 3: much improved(n=241,248) | 17 | 14
  Week 3: minimally improved(n=241,248) | 42 | 45
  Week 3: no change(n=241,248) | 146 | 165
  Week 3: minimally worse(n=241,248) | 26 | 17
  Week 3: much worse(n=241,248) | 0 | 3
  Week 4: very much improved(n=230,245) | 8 | 6
  Week 4: much improved(n=230,245) | 18 | 12
  Week 4: minimally improved(n=230,245) | 35 | 51
  Week 4: no change(n=230,245) | 152 | 154
  Week 4: minimally worse(n=230,245) | 15 | 19
  Week 4: much worse(n=230,245) | 2 | 3
  Week 5: very much improved(n=227,233) | 13 | 9
  Week 5: much improved(n=227,233) | 14 | 11
  Week 5: minimally improved(n=227,233) | 34 | 46
  Week 5: no change(n=227,233) | 146 | 151
  Week 5: minimally worse(n=227,233) | 19 | 14
  Week 5: much worse(n=227,233) | 1 | 2
  Week 6: very much improved(n=224,226) | 11 | 6
  Week 6: much improved(n=224,226) | 20 | 14
  Week 6: minimally improved(n=224,226) | 39 | 41
  Week 6: no change(n=224,226) | 139 | 148
  Week 6: minimally worse(n=224,226) | 13 | 17
  Week 6: much worse(n=224,226) | 2 | 0
  Week 7: very much improved(n=226,226) | 19 | 9
  Week 7: much improved(n=226,226) | 23 | 18
  Week 7: minimally improved(n=226,226) | 32 | 34
  Week 7: no change(n=226,226) | 136 | 150
  Week 7: minimally worse(n=226,226) | 14 | 13
  Week 7: much worse(n=226,226) | 2 | 2
  Week 8: very much improved(n=221,217) | 19 | 12
  Week 8: much improved(n=221,217) | 18 | 15
  Week 8: minimally improved(n=221,217) | 37 | 40
  Week 8: no change(n=221,217) | 131 | 139
  Week 8: minimally worse(n=221,217) | 15 | 10
  Week 8: much worse(n=221,217) | 0 | 1
  Week 8: very much worse(n=221,217) | 1 | 0
  Week 9: very much improved(n=218,214) | 19 | 13
  Week 9: much improved(n=218,214) | 19 | 16
  Week 9: minimally improved(n=218,214) | 36 | 31
  Week 9: no change(n=218,214) | 129 | 141
  Week 9: minimally worse(n=218,214) | 15 | 13
  Week 10: very much improved(n=212,211) | 20 | 13
  Week 10: much improved(n=212,211) | 21 | 18
  Week 10: minimally improved(n=212,211) | 30 | 35
  Week 10: no change(n=212,211) | 124 | 133
  Week 10: minimally worse(n=212,211) | 16 | 11
  Week 10: much worse(n=212,211) | 1 | 1
  Week 11: very much improved(n=211,205) | 23 | 15
  Week 11: much improved(n=211,205) | 17 | 14
  Week 11: minimally improved(n=211,205) | 38 | 35
  Week 11: no change(n=211,205) | 120 | 129
  Week 11: minimally worse(n=211,205) | 13 | 10
  Week 11: much worse(n=211,205) | 0 | 2
  Week 12: very much improved(n=210,204) | 19 | 17
  Week 12: much improved(n=210,204) | 19 | 13
  Week 12: minimally improved(n=210,204) | 34 | 39
  Week 12: no change(n=210,204) | 127 | 124
  Week 12: minimally worse(n=210,204) | 11 | 11
  Week 13: very much improved(n=211,200) | 18 | 16
  Week 13: much improved(n=211,200) | 19 | 13
  Week 13: minimally improved(n=211,200) | 34 | 40
  Week 13: no change(n=211,200) | 127 | 121
  Week 13: minimally worse(n=211,200) | 12 | 10
  Week 13: much worse(n=211,200) | 1 | 0
  Week 16: very much improved(n=203,199) | 17 | 15
  Week 16: much improved(n=203,199) | 27 | 16
  Week 16: minimally improved(n=203,199) | 26 | 33
  Week 16: no change(n=203,199) | 119 | 119
  Week 16: minimally worse(n=203,199) | 14 | 12
  Week 16: much worse(n=203,199) | 0 | 4
  Week 24: very much improved(n=196,193) | 17 | 13
  Week 24: much improved(n=196,193) | 17 | 18
  Week 24: minimally improved(n=196,193) | 24 | 31
  Week 24: no change(n=196,193) | 127 | 125
  Week 24: minimally worse(n=196,193) | 10 | 6
  Week 24: much worse(n=196,193) | 1 | 0
  Week 32: very much improved(n=188,188) | 15 | 19
  Week 32: much improved(n=188,188) | 19 | 21
  Week 32: minimally improved(n=188,188) | 27 | 31
  Week 32: no change(n=188,188) | 118 | 113
  Week 32: minimally worse(n=188,188) | 9 | 3
  Week 32: much worse(n=188,188) | 0 | 1
  Week 40: very much improved(n=180,182) | 10 | 17
  Week 40: much improved(n=180,182) | 23 | 15
  Week 40: minimally improved(n=180,182) | 23 | 32
  Week 40: no change(n=180,182) | 117 | 109
  Week 40: minimally worse(n=180,182) | 6 | 7
  Week 40: much worse(n=180,182) | 0 | 2
  Week 40: very much worse(n=180,182) | 1 | 0
  Week 52: very much improved(n=178,180) | 20 | 22
  Week 52: much improved(n=178,180) | 20 | 13
  Week 52: minimally improved(n=178,180) | 25 | 26
  Week 52: no change(n=178,180) | 110 | 112
  Week 52: minimally worse(n=178,180) | 3 | 7

7. Other Pre Specified Outcome: Number of Participants With Clinical Global Impression - Severity (CGI-S) Score
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 16, 24, 32, 40, 52
Population: Safety analysis population included all participants who took at least 1 dose of randomized study medication, including partial doses, and had a safety measurement. Here, the 'n' is signifying those participants who were evaluable for this measure at the specific categories for each arm group.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
participants
  Baseline:Normal; Week 1:Normal (n=250,263) | 105 | 100
  Baseline:Borderline; Week 1:Normal (n=250,263) | 7 | 8
  Baseline:Mildly; Week 1:Normal (n=250,263) | 4 | 1
  Baseline:Moderately; Week 1:Normal (n=250,263) | 1 | 0
  Baseline:Normal; Week 1:Borderline (n=250,263) | 3 | 3
  Baseline:Borderline; Week 1:Borderline (n=250,263) | 31 | 42
  Baseline:Mildly; Week 1:Borderline (n=250,263) | 9 | 3
  Baseline:Moderately; Week 1:Borderline (n=250,263) | 2 | 3
  Baseline:Normal; Week 1:Mildly (n=250,263) | 0 | 2
  Baseline:Borderline; Week 1:Mildly (n=250,263) | 4 | 1
  Baseline:Mildly; Week 1:Mildly (n=250,263) | 46 | 56
  Baseline:Moderately; Week 1:Mildly (n=250,263) | 6 | 9
  Baseline:Borderline; Week 1:Moderately (n=250,263) | 1 | 2
  Baseline:Mildly; Week 1:Moderately (n=250,263) | 1 | 0
  Baseline:Moderately; Week 1:Moderately (n=250,263) | 28 | 30
  Baseline:Markedly; Week 1:Moderately (n=250,263) | 1 | 0
  Baseline:Markedly; Week 1:Markedly (n=250,263) | 1 | 3
  Baseline:Normal; Week 2:Normal (n=244,254) | 102 | 96
  Baseline:Borderline; Week 2:Normal (n=244,254) | 13 | 12
  Baseline:Mildly; Week 2:Normal (n=244,254) | 5 | 0
  Baseline: Moderately; Week 2:Normal (n=244,254) | 0 | 1
  Baseline:Normal; Week 2:Borderline (n=244,254) | 1 | 5
  Baseline:Borderline; Week 2:Borderline (n=244,254) | 22 | 37
  Baseline:Mildly; Week 2:Borderline (n=244,254) | 10 | 7
  Baseline:Moderately; Week 2:Borderline (n=244,254) | 4 | 4
  Baseline:Normal; Week 2:Mildly (n=244,254) | 3 | 2
  Baseline:Borderline; Week 2:Mildly (n=244,254) | 4 | 0
  Baseline:Mildly; Week 2:Mildly (n=244,254) | 40 | 48
  Baseline:Moderately; Week 2:Mildly (n=244,254) | 10 | 12
  Baseline:Markedly; Week 2:Mildly (n=244,254) | 1 | 0
  Baseline:Normal; Week 2:Moderately (n=244,254) | 2 | 0
  Baseline:Borderline; Week 2:Moderately (n=244,254) | 1 | 1
  Baseline:Mildly; Week 2:Moderately (n=244,254) | 2 | 2
  Baseline:Moderately; Week 2:Moderately (n=244,254) | 20 | 24
  Baseline:Markedly; Week 2:Moderately (n=244,254) | 0 | 1
  Baseline: Moderately; Week 2:Markedly (n=244,254) | 3 | 0
  Baseline:Markedly; Week 2:Markedly (n=244,254) | 1 | 2
  Baseline:Normal; Week 3:Normal (n=241,247) | 101 | 95
  Baseline:Borderline; Week 3:Normal (n=241,247) | 18 | 16
  Baseline:Mildly; Week 3:Normal (n=241,247) | 6 | 4
  Baseline:Moderately; Week 3:Normal (n=241,247) | 2 | 0
  Baseline:Normal; Week 3:Borderline (n=241,247) | 3 | 2
  Baseline:Borderline; Week 3:Borderline (n=241,247) | 16 | 34
  Baseline:Mildly; Week 3:Borderline (n=241,247) | 8 | 7
  Baseline:Moderately; Week 3:Borderline (n=241,247) | 4 | 2
  Baseline:Normal; Week 3:Mildly (n=241,247) | 2 | 0
  Baseline:Borderline; Week 3:Mildly (n=241,247) | 6 | 2
  Baseline:Mildly; Week 3:Mildly (n=241,247) | 42 | 42
  Baseline:Moderately; Week 3:Mildly (n=241,247) | 10 | 17
  Baseline:Markedly; Week 3:Mildly (n=241,247) | 1 | 0
  Baseline:Normal; Week 3:Moderately (n=241,247) | 0 | 2
  Baseline:Mildly; Week 3:Moderately (n=241,247) | 2 | 1
  Baseline:Moderately; Week 3:Moderately (n=241,247) | 19 | 20
  Baseline:Markedly; Week 3:Moderately (n=241,247) | 0 | 1
  Baseline:Moderately; Week 3:Markedly (n=241,247) | 0 | 1
  Baseline:Markedly; Week 3:Markedly (n=241,247) | 1 | 1
  Baseline:Normal; Week 4:Normal (n=230,244) | 101 | 92
  Baseline:Borderline; Week 4:Normal (n=230,244) | 17 | 17
  Baseline:Mildly; Week 4:Normal (n=230,244) | 7 | 5
  Baseline:Moderately; Week 4:Normal (n=230,244) | 4 | 1
  Baseline:Normal; Week 4:Borderline (n=230,244) | 2 | 5
  Baseline:Borderline; Week 4:Borderline (n=230,244) | 17 | 27
  Baseline:Mildly; Week 4:Borderline (n=230,244) | 8 | 7
  Baseline:Moderately; Week 4:Borderline (n=230,244) | 1 | 3
  Baseline:Normal; Week 4:Mildly (n=230,244) | 0 | 2
  Baseline:Borderline; Week 4:Mildly (n=230,244) | 3 | 2
  Baseline:Mildly; Week 4:Mildly (n=230,244) | 39 | 43
  Baseline:Moderately; Week 4:Mildly (n=230,244) | 11 | 15
  Baseline:Markedly; Week 4:Mildly (n=230,244) | 1 | 1
  Baseline:Borderline; Week 4:Moderately (n=230,244) | 2 | 0
  Baseline:Mildly; Week 4:Moderately (n=230,244) | 2 | 2
  Baseline:Moderately; Week 4:Moderately (n=230,244) | 12 | 2
  Baseline:Markedly; Week 4:Moderately (n=230,244) | 1 | 18
  Baseline:Borderline; Week 4:Markedly (n=230,244) | 1 | 0
  Baseline:Moderately; Week 4:Markedly (n=230,244) | 1 | 0
  Baseline:Markedly; Week 4:Markedly (n=230,244) | 0 | 2
  Baseline:Normal; Week 5:Normal (n=227,232) | 98 | 88
  Baseline:Borderline; Week 5:Normal (n=227,232) | 19 | 16
  Baseline:Mildly; Week 5:Normal (n=227,232) | 8 | 6
  Baseline:Moderately; Week 5:Normal (n=227,232) | 4 | 4
  Baseline:Normal; Week 5:Borderline (n=227,232) | 2 | 1
  Baseline:Borderline; Week 5:Borderline (n=227,232) | 13 | 30
  Baseline:Mildly; Week 5:Borderline (n=227,232) | 8 | 4
  Baseline:Moderately; Week 5:Borderline (n=227,232) | 2 | 3
  Baseline:Normal; Week 5:Mildly (n=227,232) | 2 | 1
  Baseline:Borderline; Week 5:Mildly (n=227,232) | 6 | 2
  Baseline:Mildly; Week 5:Mildly (n=227,232) | 36 | 39
  Baseline:Moderately; Week 5:Mildly (n=227,232) | 11 | 15
  Baseline:Markedly; Week 5:Mildly (n=227,232) | 2 | 1
  Baseline:Normal; Week 5:Moderately (n=227,232) | 0 | 1
  Baseline:Borderline; Week 5:Moderately (n=227,232) | 1 | 0
  Baseline:Mildly; Week 5:Moderately (n=227,232) | 2 | 4
  Baseline:Moderately; Week 5:Moderately (n=227,232) | 12 | 15
  Baseline:Markedly; Week 5:Moderately (n=227,232) | 0 | 1
  Baseline:Moderately; Week 5:Markedly (n=227,232) | 1 | 1
  Baseline:Normal; Week 6:Normal (n=224,225) | 96 | 84
  Baseline:Borderline; Week 6:Normal (n=224,225) | 22 | 18
  Baseline:Mildly; Week 6:Normal (n=224,225) | 10 | 4
  Baseline:Moderately; Week 6:Normal (n=224,225) | 3 | 1
  Baseline:Normal; Week 6:Borderline (n=224,225) | 3 | 3
  Baseline:Borderline; Week 6:Borderline (n=224,225) | 11 | 24
  Baseline:Mildly; Week 6:Borderline (n=224,225) | 6 | 7
  Baseline:Moderately; Week 6:Borderline (n=224,225) | 5 | 4
  Baseline:Normal; Week 6:Mildly (n=224,225) | 2 | 2
  Baseline:Borderline; Week 6:Mildly (n=224,225) | 5 | 2
  Baseline:Mildly; Week 6:Mildly (n=224,225) | 38 | 37
  Baseline:Moderately; Week 6:Mildly (n=224,225) | 8 | 15
  Baseline:Markedly; Week 6:Mildly (n=224,225) | 2 | 1
  Baseline:Normal; Week 6:Moderately (n=224,225) | 0 | 3
  Baseline:Borderline; Week 6:Moderately (n=224,225) | 1 | 1
  Baseline:Mildly; Week 6:Moderately (n=224,225) | 1 | 3
  Baseline:Moderately; Week 6:Moderately (n=224,225) | 10 | 14
  Baseline:Moderately; Week 6:Markedly (n=224,225) | 1 | 1
  Baseline:Markedly; Week 6:Markedly (n=224,225) | 0 | 1
  Baseline:Normal; Week 7:Normal (n=226,225) | 93 | 88
  Baseline:Borderline; Week 7:Normal (n=226,225) | 23 | 20
  Baseline:Mildly; Week 7:Normal (n=226,225) | 14 | 5
  Baseline:Moderately; Week 7:Normal (n=226,225) | 3 | 1
  Baseline:Normal; Week 7:Borderline (n=226,225) | 5 | 2
  Baseline:Borderline; Week 7:Borderline (n=226,225) | 13 | 23
  Baseline:Mildly; Week 7:Borderline (n=226,225) | 4 | 6
  Baseline:Moderately; Week 7:Borderline (n=226,225) | 5 | 8
  Baseline:Markedly; Week 7:Borderline (n=226,225) | 1 | 0
  Baseline:Normal; Week 7:Mildly (n=226,225) | 2 | 0
  Baseline:Borderline; Week 7:Mildly (n=226,225) | 2 | 2
  Baseline:Mildly; Week 7:Mildly (n=226,225) | 36 | 37
  Baseline:Moderately; Week 7:Mildly (n=226,225) | 10 | 10
  Baseline:Markedly; Week 7:Mildly (n=226,225) | 1 | 1
  Baseline:Normal; Week 7:Moderately (n=226,225) | 0 | 1
  Baseline:Borderline; Week 7:Moderately (n=226,225) | 1 | 1
  Baseline:Mildly; Week 7:Moderately (n=226,225) | 2 | 4
  Baseline:Moderately; Week 7:Moderately (n=226,225) | 10 | 14
  Baseline:Markedly; Week 7:Moderately (n=226,225) | 0 | 1
  Baseline:Moderately; Week 7:Markedly (n=226,225) | 1 | 1
  Baseline:Normal; Week 8:Normal (n=221,216) | 92 | 87
  Baseline:Borderline; Week 8:Normal (n=221,216) | 21 | 19
  Baseline:Mildly; Week 8:Normal (n=221,216) | 12 | 6
  Baseline:Moderately; Week 8:Normal (n=221,216) | 3 | 3
  Baseline:Normal; Week 8:Borderline (n=221,216) | 4 | 2
  Baseline:Borderline; Week 8:Borderline (n=221,216) | 14 | 19
  Baseline:Mildly; Week 8:Borderline (n=221,216) | 6 | 7
  Baseline:Moderately; Week 8:Borderline (n=221,216) | 7 | 5
  Baseline:Markedly; Week 8:Borderline (n=221,216) | 2 | 0
  Baseline:Normal; Week 8:Mildly (n=221,216) | 2 | 0
  Baseline:Borderline; Week 8:Mildly (n=221,216) | 3 | 2
  Baseline:Mildly; Week 8:Mildly (n=221,216) | 32 | 35
  Baseline:Moderately; Week 8:Mildly (n=221,216) | 9 | 13
  Baseline:Markedly; Week 8:Mildly (n=221,216) | 0 | 1
  Baseline:Normal; Week 8:Moderately (n=221,216) | 1 | 0
  Baseline:Mildly; Week 8:Moderately (n=221,216) | 3 | 3
  Baseline:Moderately; Week 8:Moderately (n=221,216) | 9 | 12
  Baseline:Markedly; Week 8:Moderately (n=221,216) | 0 | 1
  Baseline:Mildly; Week 8:Markedly (n=221,216) | 0 | 1
  Baseline:Moderately; Week 8:Markedly (n=221,216) | 1 | 0
  Baseline:Normal; Week 9:Normal (n=218,213) | 91 | 87
  Baseline:Borderline; Week 9:Normal (n=218,213) | 22 | 18
  Baseline:Mildly; Week 9:Normal (n=218,213) | 11 | 5
  Baseline:Moderately; Week 9:Normal (n=218,213) | 4 | 4
  Baseline:Normal; Week 9:Borderline (n=218,213) | 3 | 2
  Baseline:Borderline; Week 9:Borderline (n=218,213) | 13 | 19
  Baseline:Mildly; Week 9:Borderline (n=218,213) | 6 | 3
  Baseline:Moderately; Week 9:Borderline (n=218,213) | 6 | 8
  Baseline:Markedly; Week 9:Borderline (n=218,213) | 2 | 1
  Baseline:Normal; Week 9:Mildly (n=218,213) | 3 | 0
  Baseline:Borderline; Week 9:Mildly (n=218,213) | 2 | 4
  Baseline:Mildly; Week 9:Mildly (n=218,213) | 34 | 38
  Baseline:Moderately; Week 9:Mildly (n=218,213) | 10 | 9
  Baseline:Mildly; Week 9:Moderately (n=218,213) | 1 | 0
  Baseline:Moderately; Week 9:Moderately (n=218,213) | 8 | 12
  Baseline:Markedly; Week 9:Moderately (n=218,213) | 0 | 1
  Baseline:Mildly; Week 9:Markedly (n=218,213) | 1 | 1
  Baseline:Moderately; Week 9:Markedly (n=218,213) | 1 | 1
  Baseline:Normal; Week 10:Normal (n=212,210) | 88 | 85
  Baseline:Borderline; Week 10:Normal (n=212,210) | 20 | 21
  Baseline:Mildly; Week 10:Normal (n=212,210) | 13 | 5
  Baseline:Moderately; Week 10:Normal (n=212,210) | 7 | 5
  Baseline:Normal; Week 10:Borderline (n=212,210) | 5 | 1
  Baseline:Borderline; Week 10:Borderline (n=212,210 | 14 | 18
  Baseline:Mildly; Week 10:Borderline (n=212,210) | 6 | 6
  Baseline:Moderately; Week 10:Borderline(n=212,210) | 4 | 7
  Baseline:Markedly; Week 10:Borderline(n=212,210) | 2 | 1
  Baseline:Normal; Week 10:Mildly (n=212,210) | 1 | 1
  Baseline:Borderline; Week 10:Mildly (n=212,210) | 1 | 2
  Baseline:Mildly; Week 10:Mildly (n=212,210) | 29 | 35
  Baseline:Moderately; Week 10:Mildly (n=212,210) | 8 | 11
  Baseline:Normal; Week 10:Moderately (n=212,210) | 1 | 0
  Baseline:Mildly; Week 10:Moderately (n=212,210) | 3 | 1
  Baseline:Moderately; Week 10:Moderately(n=212,210) | 9 | 9
  Baseline:Markedly; Week 10:Moderately (n=212,210) | 0 | 1
  Baseline:Moderately; Week 10:Markedly (n=212,210) | 1 | 1
  Baseline:Normal; Week 11:Normal (n=211,205) | 90 | 81
  Baseline:Borderline; Week 11:Normal (n=211,205) | 23 | 22
  Baseline:Mildly; Week 11:Normal (n=211,205) | 13 | 6
  Baseline:Moderately; Week 11:Normal (n=211,205) | 7 | 5
  Baseline:Markedly; Week 11:Normal (n=211,205) | 1 | 0
  Baseline:Normal; Week 11:Borderline (n=211,205) | 3 | 2
  Baseline:Borderline; Week 11:Borderline(n=211,205) | 10 | 15
  Baseline:Mildly; Week 11:Borderline (n=211,205) | 6 | 3
  Baseline:Moderately; Week 11:Borderline(n=211,205) | 3 | 6
  Baseline:Markedly; Week 11:Borderline (n=211,205) | 1 | 1
  Baseline:Normal; Week 11:Mildly (n=211,205) | 1 | 0
  Baseline:Borderline; Week 11:Mildly (n=211,205) | 2 | 3
  Baseline:Mildly; Week 11:Mildly (n=211,205) | 30 | 34
  Baseline:Moderately; Week 11:Mildly (n=211,205) | 9 | 13
  Baseline:Normal; Week 11:Moderately (n=211,205) | 0 | 1
  Baseline:Mildly; Week 11:Moderately (n=211,205) | 3 | 1
  Baseline:Moderately; Week 11:Moderately(n=211,205) | 8 | 10
  Baseline:Markedly; Week 11:Moderately (n=211,205) | 0 | 1
  Baseline:Mildly; Week 11:Markedly (n=211,205) | 0 | 1
  Baseline:Normal; Week 12:Normal (n=210,203) | 89 | 79
  Baseline:Borderline; Week 12:Normal (n=210,203) | 23 | 22
  Baseline:Mildly; Week 12:Normal (n=210,203) | 13 | 6
  Baseline:Moderately; Week 12:Normal (n=210,203) | 6 | 8
  Baseline:Markedly; Week 12:Normal (n=210,203) | 1 | 0
  Baseline:Normal; Week 12:Borderline (n=210,203) | 4 | 2
  Baseline:Borderline; Week 12:Borderline(n=210,203) | 12 | 16
  Baseline:Mildly; Week 12:Borderline (n=210,203) | 6 | 4
  Baseline:Moderately; Week 12:Borderline(n=210,203) | 4 | 3
  Baseline:Markedly; Week 12:Borderline (n=210,203) | 1 | 1
  Baseline:Normal; Week 12:Mildly (n=210,203) | 0 | 2
  Baseline:Borderline; Week 12:Mildly (n=210,203) | 0 | 1
  Baseline:Mildly; Week 12:Mildly (n=210,203) | 30 | 34
  Baseline:Moderately; Week 12:Mildly (n=210,203) | 9 | 14
  Baseline:Borderline; Week 12:Moderately(n=210,203) | 0 | 1
  Baseline:Mildly; Week 12:Moderately (n=210,203) | 3 | 3
  Baseline:Moderately; Week 12:Moderately(n=210,203) | 8 | 6
  Baseline:Markedly; Week 12:Moderately(n=210,203) | 0 | 1
  Baseline:Moderately; Week 12:Markedly(n=210,203) | 1 | 0
  Baseline:Normal; Week 13:Normal (n=211,199) | 92 | 78
  Baseline:Borderline; Week 13:Normal (n=211,199) | 22 | 21
  Baseline:Mildly; Week 13:Normal (n=211,199) | 13 | 5
  Baseline:Moderately; Week 13:Normal (n=211,199) | 6 | 9
  Baseline:Markedly; Week 13:Normal (n=211,199) | 2 | 0
  Baseline:Normal; Week 13:Borderline (n=211,199) | 3 | 3
  Baseline:Borderline; Week 13:Borderline(n=211,199) | 11 | 17
  Baseline:Mildly; Week 13:Borderline (n=211,199) | 7 | 6
  Baseline:Moderately; Week 13:Borderline(n=211,199) | 5 | 4
  Baseline:Markedly; Week 13:Borderline(n=211,199) | 0 | 1
  Baseline:Borderline; Week 13:Mildly (n=211,199) | 0 | 3
  Baseline:Mildly; Week 13:Mildly (n=211,199) | 30 | 32
  Baseline:Moderately; Week 13:Mildly (n=211,199) | 9 | 11
  Baseline:Mildly; Week 13:Moderately (n=211,199) | 3 | 1
  Baseline:Moderately; Week 13:Moderately(n=211,199) | 7 | 7
  Baseline:Markedly; Week 13:Moderately(n=211,199) | 0 | 1
  Baseline:Moderately; Week 13:Markedly (n=211,199) | 1 | 0
  Baseline:Normal; Week 16:Normal (n=203,198) | 91 | 78
  Baseline:Borderline; Week 16:Normal (n=203,198) | 19 | 20
  Baseline:Mildly; Week 16:Normal (n=203,198) | 14 | 6
  Baseline:Moderately; Week 16:Normal (n=203,198) | 7 | 11
  Baseline:Markedly; Week 16:Normal (n=203,198) | 2 | 0
  Baseline:Normal; Week 16:Borderline (n=203,198) | 2 | 2
  Baseline:Borderline; Week 16:Borderline(n=203,198) | 11 | 16
  Baseline:Mildly; Week 16:Borderline (n=203,198) | 4 | 5
  Baseline:Moderately; Week 16:Borderline(n=203,198) | 2 | 2
  Baseline:Markedly; Week 16:Borderline (n=203,198) | 0 | 1
  Baseline:Normal; Week 16:Mildly (n=203,198) | 1 | 2
  Baseline:Borderline; Week 16:Mildly (n=203,198) | 0 | 3
  Baseline:Mildly; Week 16:Mildly (n=203,198) | 30 | 30
  Baseline:Moderately; Week 16:Mildly (n=203,198) | 11 | 8
  Baseline:Borderline; Week 16:Moderately(n=203,198) | 0 | 2
  Baseline:Mildly; Week 16:Moderately (n=203,198) | 3 | 2
  Baseline:Moderately; Week 16:Moderately(n=203,198) | 4 | 8
  Baseline:Markedly; Week 16:Moderately (n=203,198) | 0 | 1
  Baseline:Moderately; Week 16:Markedly (n=203,198) | 2 | 1
  Baseline:Normal; Week 24:Normal (n=196,192) | 88 | 78
  Baseline:Borderline; Week 24:Normal (n=196,192) | 18 | 19
  Baseline:Mildly; Week 24:Normal (n=196,192) | 15 | 6
  Baseline:Moderately; Week 24:Normal (n=196,192) | 5 | 8
  Baseline:Markedly; Week 24:Normal (n=196,192) | 2 | 0
  Baseline:Normal; Week 24:Borderline (n=196,192) | 0 | 3
  Baseline:Borderline; Week 24:Borderline(n=196,192) | 13 | 14
  Baseline:Mildly; Week 24:Borderline (n=196,192) | 4 | 6
  Baseline:Moderately; Week 24:Borderline(n=196,192) | 2 | 2
  Baseline:Markedly; Week 24:Borderline (n=196,192) | 0 | 1
  Baseline:Normal; Week 24:Mildly (n=196,192) | 2 | 1
  Baseline:Borderline; Week 24:Mildly (n=196,192) | 0 | 3
  Baseline:Mildly; Week 24:Mildly (n=196,192) | 27 | 31
  Baseline:Moderately; Week 24:Mildly (n=196,192) | 8 | 12
  Baseline:Mildly; Week 24:Moderately (n=196,192) | 4 | 0
  Baseline:Moderately; Week 24:Moderately(n=196,192) | 7 | 7
  Baseline:Markedly; Week 24:Moderately (n=196,192) | 0 | 1
  Baseline:Moderately; Week 24:Markedly (n=196,192) | 1 | 0
  Baseline:Normal; Week 32:Normal (n=188,187) | 82 | 77
  Baseline:Borderline; Week 32:Normal (n=188,187) | 16 | 20
  Baseline:Mildly; Week 32:Normal (n=188,187) | 10 | 8
  Baseline:Moderately; Week 32:Normal (n=188,187) | 4 | 9
  Baseline:Markedly; Week 32:Normal (n=188,187) | 2 | 0
  Baseline:Normal; Week 32:Borderline (n=188,187) | 0 | 1
  Baseline:Borderline; Week 32:Borderline(n=188,187) | 12 | 15
  Baseline:Mildly; Week 32:Borderline (n=188,187) | 9 | 7
  Baseline:Moderately; Week 32:Borderline(n=188,187) | 4 | 1
  Baseline:Markedly; Week 32:Borderline (n=188,187) | 0 | 1
  Baseline:Normal; Week 32:Mildly (n=188,187) | 2 | 0
  Baseline:Borderline; Week 32:Mildly (n=188,187) | 0 | 1
  Baseline:Mildly; Week 32:Mildly (n=188,187) | 28 | 29
  Baseline:Moderately; Week 32:Mildly (n=188,187) | 8 | 11
  Baseline:Markedly; Week 32:Mildly (n=188,187) | 0 | 1
  Baseline:Mildly; Week 32:Moderately (n=188,187) | 3 | 0
  Baseline:Moderately; Week 32:Moderately(n=188,187) | 7 | 5
  Baseline:Borderline; Week 32:Markedly (n=188,187) | 0 | 1
  Baseline:Moderately; Week 32:Markedly (n=188,187) | 1 | 0
  Baseline:Normal; Week 40:Normal (n=180,181) | 81 | 71
  Baseline:Borderline; Week 40:Normal (n=180,181) | 17 | 20
  Baseline:Mildly; Week 40:Normal (n=180,181) | 11 | 7
  Baseline:Moderately; Week 40:Normal (n=180,181) | 2 | 7
  Baseline:Markedly; Week 40:Normal (n=180,181) | 2 | 0
  Baseline:Normal; Week 40:Borderline (n=180,181) | 0 | 2
  Baseline:Borderline; Week 40:Borderline(n=180,181) | 9 | 15
  Baseline:Mildly; Week 40:Borderline (n=180,181) | 8 | 6
  Baseline:Moderately; Week 40:Borderline(n=180,181) | 4 | 2
  Baseline:Markedly; Week 40:Borderline (n=180,181) | 0 | 1
  Baseline:Normal; Week 40:Mildly (n=180,181) | 1 | 0
  Baseline:Borderline; Week 40:Mildly (n=180,181) | 2 | 2
  Baseline:Mildly; Week 40:Mildly (n=180,181) | 25 | 28
  Baseline:Moderately; Week 40:Mildly (n=180,181) | 11 | 12
  Baseline:Markedly; Week 40:Mildly (n=180,181) | 0 | 1
  Baseline:Normal; Week 40:Moderately (n=180,181) | 0 | 1
  Baseline:Mildly; Week 40:Moderately (n=180,181) | 2 | 1
  Baseline:Moderately; Week 40:Moderately(n=180,181) | 4 | 3
  Baseline:Moderately; Week 40:Markedly (n=180,181) | 1 | 2
  Baseline:Normal; Week 52:Normal (n=178,179) | 81 | 69
  Baseline:Borderline; Week 52:Normal (n=178,179) | 19 | 20
  Baseline:Mildly; Week 52:Normal (n=178,179) | 12 | 7
  Baseline:Moderately; Week 52:Normal (n=178,179) | 4 | 7
  Baseline:Markedly; Week 52:Normal (n=178,179) | 2 | 0
  Baseline:Normal; Week 52:Borderline (n=178,179) | 1 | 4
  Baseline:Borderline; Week 52:Borderline(n=178,179) | 8 | 14
  Baseline:Mildly; Week 52:Borderline (n=178,179) | 8 | 8
  Baseline:Moderately; Week 52:Borderline(n=178,179) | 4 | 4
  Baseline:Markedly; Week 52:Borderline (n=178,179) | 0 | 1
  Baseline:Normal; Week 52:Mildly (n=178,179) | 1 | 0
  Baseline:Borderline; Week 52:Mildly (n=178,179) | 0 | 2
  Baseline:Mildly; Week 52:Mildly (n=178,179) | 24 | 26
  Baseline:Moderately; Week 52:Mildly (n=178,179) | 8 | 11
  Baseline:Mildly; Week 52:Moderately (n=178,179) | 1 | 1
  Baseline:Moderately; Week 52:Moderately(n=178,179) | 4 | 4
  Baseline:Markedly; Week 52:Moderately (n=178,179) | 0 | 1
  Baseline:Moderately; Week 52:Markedly (n=178,179) | 1 | 0

8. Other Pre Specified Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) - Total Score
Description: Measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Change: mean score at observation minus mean score at baseline.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 16
Population: Safety analysis population included all participants who took at least 1 dose of randomized study medication, including partial doses, and had a safety measurement. 'n' is signifying those participants who were evaluated for this measure at the satisfaction level for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
Units on a scale
  Baseline(n=256,269) | 7.6 (7.38) | 7.9 (7.51)
  Change at Week 1(n=250,265) | -1.2 (3.95) | -0.6 (4.17)
  Change at Week 2(n= 245, 255) | -1.0 (6.06) | -1.1 (5.33)
  Change at Week 3(n= 241, 249) | -1.9 (5.19) | -1.8 (4.96)
  Change at Week 4(n= 230, 246) | -2.2 (5.62) | -1.5 (5.96)
  Change at Week 5(n=228, 235) | -2.1 (6.01) | -2.3 (6.09)
  Change at Week 6(n=224, 227) | -2.2 (6.15) | -2.3 (5.84)
  Change at Week 7(n=226, 227) | -2.3 (6.57) | -2.4 (5.94)
  Change at Week 8(n=221, 218) | -2.7 (6.51) | -2.6 (6.02)
  Change at Week 9(n=218, 216) | -2.9 (6.11) | -2.5 (6.55)
  Change at Week 10(n=214, 212) | -2.9 (6.21) | -2.8 (6.15)
  Change at Week 11(n= 211, 206) | -3.2 (6.30) | -2.9 (6.13)
  Change at Week 12(n= 210, 205) | -3.4 (6.20) | -3.2 (6.34)
  Change at Week 13(n= 211, 201) | -3.0 (6.39) | -3.6 (5.88)
  Change at Week 16(n= 202, 197) | -3.1 (6.36) | -3.2 (6.61)

9. Other Pre Specified Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) - Total Score
Description: HAM-A measures treatment-related changes in generalized anxiety symptoms; 14 item questionnaire scored 0 (not present) to 4 (very severe); possible range 0 to 56. Lower score indicates less affected. Change: mean score at observation minus mean score at baseline.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
Units on a scale
  Baseline(n=256,269) | 6.1 (5.23) | 6.4 (5.17)
  Change at Week 1(n=250,265) | -0.5 (2.54) | -0.7 (3.15)
  Change at Week 2(n= 245, 255) | -0.7 (3.98) | -0.5 (3.79)
  Change at Week 3(n= 241, 249) | -1.3 (3.41) | -1.2 (3.68)
  Change at Week 4(n= 230, 246) | -1.6 (3.72) | -1.2 (3.87)
  Change at Week 5(n=228, 235) | -1.6 (4.05) | -1.6 (4.00)
  Change at Week 6(n=224, 227) | -1.7 (4.03) | -1.6 (4.00)
  Change at Week 7(n=226, 227) | -2.0 (4.40) | -1.8 (4.32)
  Change at Week 8(n=221, 218) | -1.9 (4.65) | -1.9 (4.10)
  Change at Week 9(n=218, 216) | -2.0 (4.40) | -1.9 (3.94)
  Change at Week 10(n=214, 212) | -2.2 (4.24) | -2.0 (4.12)
  Change at Week 11(n= 211, 206) | -2.3 (4.48) | -2.1 (4.31)
  Change at Week 12(n= 210, 205) | -2.3 (4.27) | -2.4 (4.47)
  Change at Week 13(n= 211, 201) | -2.4 (4.49) | -2.7 (4.34)
  Change at Week 16(n= 202, 197) | -2.7 (4.67) | -2.5 (4.28)

10. Other Pre Specified Outcome: Change From Baseline in Barratt Impulsiveness Scale (BIS-11) - Total Score
Description: The BIS-11 is a self-administered 30 items questionnaire to assess measure of impulsivity. Items are scored on a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/always). Total score range from 30 to 120. Barratt suggested that a total score of greater than or equal to 75 could indicate an impulse-control disorder, whereas a total score in the range of 70 to 75 could indicate pathological impulsivity.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
Units on a scale
  Baseline(n=256,269) | 65.1 (6.42) | 64.2 (7.30)
  Change at Week 1(n=250,265) | -0.5 (4.36) | -0.8 (4.26)
  Change at Week 2(n= 244, 255) | -0.8 (4.73) | -1.1 (4.83)
  Change at Week 3(n= 241, 249) | -1.0 (4.75) | -1.3 (4.81)
  Change at Week 4(n= 230, 246) | -1.0 (5.19) | -1.2 (4.95)
  Change at Week 5(n=228, 234) | -1.1 (5.27) | -1.1 (5.39)
  Change at Week 6(n=224, 226) | -1.4 (5.28) | -1.2 (5.43)
  Change at Week 7(n=226, 227) | -1.6 (5.62) | -1.3 (6.08)
  Change at Week 8(n=219, 216) | -1.3 (5.81) | -1.2 (6.54)
  Change at Week 9(n=218, 215) | -1.5 (6.25) | -1.4 (6.24)
  Change at Week 10(n=214, 211) | -1.5 (6.13) | -1.7 (6.94)
  Change at Week 11(n= 211, 205) | -1.6 (6.24) | -1.5 (6.78)
  Change at Week 12(n= 210, 204) | -1.0 (6.55) | -1.4 (7.31)
  Change at Week 13(n= 211, 201) | -1.4 (6.52) | -1.1 (7.00)
  Change at Week 16(n= 202, 196) | -1.4 (6.25) | -1.3 (6.85)

11. Other Pre Specified Outcome: Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS assessed if participant experienced following: completed suicide (1), suicide attempt (2)(response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4)("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has participant engaged in non-suicidal self-injurious behavior").
Time Frame: Baseline, Week 1 up to 30 days after Week 12 (treatment-emergent [TE]), thereafter up to Week 52 (follow-up [FU])
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 256 | 269
participants
  Baseline,Suicidal Behavior or/and Ideation | 6 | 1
  Baseline,4 | 6 | 1
  Baseline,4: wish to be dead | 6 | 1
  TE,Suicidal Behavior or/and Ideation | 15 | 20
  TE,2 | 0 | 1
  TE,4 | 15 | 19
  TE,4: wish to be dead | 15 | 18
  TE,4: non-specific active suicidal thoughts | 4 | 7
  TE,4: with any methods,without intent to act | 2 | 5
  TE,4: with some intent,without specific plan. | 0 | 3
  TE,4: with specific plan and intent | 0 | 1
  FU,Suicidal Behavior or/and Ideation | 13 | 12
  FU,1 | 1 | 0
  FU,4 | 12 | 12
  FU,4: wish to be dead | 11 | 12
  FU,4: non-specific active suicidal thoughts | 5 | 3
  FU,4: with any methods,without intent to act | 2 | 2
  FU,4: with some intent,without specific plan | 1 | 1
  FU,7 | 1 | 1

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 7/256 | 7/269
Other Adverse Events (participants affected / at risk) | 158/256 | 126/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=256) | Placebo (N=269)
Palpitations (Cardiac disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Device dislocation (General disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Ligament laxity (Musculoskeletal and connective tissue disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Depression suicidal (Psychiatric disorders) | 1 | 1
Intentional sefl-injury (Psychiatric disorders) | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Claculus ureteric (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemodynamic instability (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=256) | Placebo (N=269)
Constipation (Gastrointestinal disorders) | 15 | 9
Diarrhoea (Gastrointestinal disorders) | 16 | 12
Dry mouth (Gastrointestinal disorders) | 17 | 14
Nausea (Gastrointestinal disorders) | 69 | 28
Vomiting (Gastrointestinal disorders) | 13 | 9
Irritability (General disorders) | 28 | 22
Nasopharyngitis (Infections and infestations) | 14 | 13
Upper respiratory tract infection (Infections and infestations) | 15 | 13
Weight increased (Investigations) | 14 | 5
Headache (Nervous system disorders) | 43 | 30
Abnormal dreams (Psychiatric disorders) | 29 | 22
Agitation (Psychiatric disorders) | 17 | 10
Anxiety (Psychiatric disorders) | 18 | 25
Depression (Psychiatric disorders) | 17 | 13
Insomnia (Psychiatric disorders) | 28 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.